CLINICAL TRIAL: NCT02354937
Title: A Phase I, Open-Label, Parallel-Group Study to Evaluate the Pharmacokinetics and Safety of GSK1265744 in Subjects With Severe Renal Impairment and Healthy Matched Control Subjects
Brief Title: Pharmacokinetics Study of GSK1265744 in Subjects With Severe Renal Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 201480
Record Dates: First submitted 2015-01-29; First posted 2015-02-03 (Estimated); Last update posted 2020-08-28 (Actual); Status verified 2020-08

CONDITIONS: Infection, Human Immunodeficiency Virus; HIV Infections
Keywords: Pharmacokinetics; GSK1265744; Severe Renal Impairment
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome; HIV Infections; Renal Insufficiency | interventions — cabotegravir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Subjects with renal impairment (Experimental): Subjects with severe renal impairment will receive single oral dose of 744 30 mg
  Interventions: Drug: GSK1265744 30 mg
- Subjects with normal renal function (Active Comparator): Subjects with normal renal function will receive single oral dose of 744 30 mg
  Interventions: Drug: GSK1265744 30 mg

INTERVENTIONS:
Drug: GSK1265744 30 mg — White to almost white coated oval tablets with unit dose strength of 30 mg for oral administrations.

SUMMARY:
GSK1265744 (744) is an integrase strand transfer inhibitor (INSTI) currently in development for both the treatment and prevention of human immunodeficiency virus (HIV) infection. Renal elimination of unchanged 744 is extremely low, with no parent 744 detected in the urine after a single 30 mg radiolabeled dose. Despite the minimal contribution of renal clearance on overall 744 elimination, renal impairment may potentially inhibit some pathways of hepatic and gut drug metabolism and transport, and as a result may impact 744 pharmacokinetics. The current Food and Drug Administration (FDA) draft guidance for renal impairment studies suggests that a pharmacokinetic (PK) study in patients with renal impairment be conducted even for those drugs primarily metabolized or secreted in bile.

The study will be comprised of two cohorts (severe renal impairment and normal renal function) of 8 subjects each. Upon enrolment, each subject will be admitted to the study center and undergo serial PK sampling following a single dose of oral 744 30 milligrams (mg). Subjects will return to the clinic for follow-up evaluations 10-14 days after the 744 30 mg dose.

ELIGIBILITY:
Inclusion Criteria:

For Renally Impaired Subjects (Cohort 1)

* Between 18 and 70 years of age inclusive, at the time of signing the informed consent.
* Severe renal impairment, defined as individuals with a creatinine clearance of < 30 milliliter (mL)/minute (min) as determined by a 24-hour urine creatinine clearance done at screening.
* Renally impaired subjects must have clinical laboratory test results that are considered clinically stable in the opinion of the principal investigator. Subjects with laboratory parameters outside the reference range may be included if, in the opinion of the investigator and medical monitor, these findings will not interfere with the study or introduce additional safety risk to the subject.
* Body weight >= 50 kilograms (kg) and body mass index (BMI) within the range 19 - 38 kg/ meter (m)^2 (inclusive)
* Male or female A female subject is eligible to participate if she is not pregnant (as confirmed by a negative serum hCG test), not lactating. Women of child-bearing potential must be willing to practice acceptable methods of birth control. Pre-menopausal females defined as 12 months of spontaneous amenorrhea with one of the following: Documented tubal ligation, hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion, Hysterectomy, Bilateral Oophorectomy. Postmenopausal
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the consent form and in this protocol.

For Healthy Subjects (Cohort 2)

* Healthy control subjects will be matched for age +/-10 years to subjects in the renal impairment cohort but must also remain in the age range:

Between 18 and 70 years of age inclusive, at the time of signing the informed consent.

* Healthy as determined by the investigator or medically qualified designee based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring.
* Healthy subjects are defined as individuals with a creatinine clearance >= 90 mL/min as determined by a 24-hour urine creatinine clearance done at screening.
* Healthy control subjects will be matched for BMI +/- 25% to subjects in the renal impairment cohort but must also remain in the range of:

Body weight >=50 kg and BMI within the range 19 - 38 kg/m^2 (inclusive)

* Male or female A female subject is eligible to participate if she is not pregnant (as confirmed by a negative serum hCG test), not lactating. Women of child-bearing potential must be willing to practice acceptable methods of birth control. Pre-menopausal females defined as 12 months of spontaneous amenorrhea with one of the following: Documented tubal ligation, hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion, Hysterectomy, Bilateral Oophorectomy. Postmenopausal
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the consent form and in this protocol.

Exclusion Criteria:

For Renally Impaired Subjects (Cohort 1)

* Alanine aminotransferase (ALT) and bilirubin >1.5x upper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Current or chronic history of liver disease (including acute or chronic hepatitis B and C), or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Corrected QT Interval (QTc) > 480 millisecond (msec)

NOTES:

The QTc is the QT interval corrected for heart rate according to Fridericia's formula (QTcF) machine-read or manually over-read.

For purposes of data analysis, QT interval corrected for heart rate according to Bazette's formula (QTcB), QTcF, or a composite of available values of QTc will be used as specified in the Reporting and Analysis Plan (RAP).

* Systolic blood pressure outside the range of 90-160mmHg, or diastolic blood pressure outside the range of 45-95 millimeter of mercury (mmHg), or heart rate outside the range of 50-100 beats per minute (bpm) for female subjects or 45-100 bpm for male subjects in the presence (or absence) of stabilized antihypertensive treatment.
* Evidence of previous myocardial infarction in the past 12 months or any clinically significant active cardiovascular disease that, in the opinion of the investigator, could interfere with the safety of the subject.
* Any clinically significant conduction abnormality (not including left or right complete bundle branch block) such as atrioventricular (AV) block [Mobitz type 2 second degree or higher AV block], Wolf Parkinson White [WPW] syndrome or other aberrant pathways.
* Sinus Pauses >3 seconds.
* Any significant arrhythmia which, in the opinion of the principal investigator and GSK medical monitor, will interfere with the safety of the individual subject.
* Non-sustained or sustained ventricular tachycardia (>=3 consecutive ventricular ectopic beats).
* Signs of active infection that in the opinion of the investigator would interfere with the completion of study procedures or the safety of the subject.
* Fluctuating or rapidly deteriorating renal function, or currently receiving hemodialysis, peritoneal dialysis, or any other renal replacement therapy or other medical procedure that serves as a surrogate for renal function. Assessment of the stability of the subject's renal function will be determined by the investigator.
* History of renal transplant.
* History of inflammatory bowel disease.
* History of cholecystectomy or other gastrointestinal surgery (except appendectomy more than three months prior to study).
* History of peptic ulceration or pancreatitis within the preceding 6 months of screening.
* Any other medical condition (except renal impairment) which, in the judgment of the investigator and medical monitor, could jeopardize the integrity of the data derived from that subject or the safety of the subject. This includes but is not limited to any pre-existing condition that interferes with normal gastrointestinal anatomy or motility that could interfere with the absorption, metabolism, and/or excretion of the study drug.
* The use of any concurrent prohibited medications
* Subjects with a change in dose regimen of medically required medication within the 2 weeks prior to dosing.
* History of regular alcohol consumption within 6 months of the study defined as:

An average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 grams (g) of alcohol: 12 ounces (360 millilitre [mL]) of beer, 5 ounces (150 mL) of wine or 1.5 ounces (45 mL) of 80 proof distilled spirits.

* Inability or unwillingness to comply with lifestyle and/or dietary restrictions
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation. In addition, if heparin is used during PK sampling, subjects with a history of sensitivity to heparin or heparin-induced thrombocytopenia should not be enrolled.
* A pre-study screen positive for alcohol, cocaine, amphetamines, phencyclidine (PCP), and/or barbiturates. A positive drug screen is permitted if it is due to a prescribed medication, provided that medication is not a Prohibited Medication.
* A positive test for HIV antibody.
* A creatinine clearance <15 mL/min as determined by 24-hour urine collection.
* A clinically significant elevation in serum potassium at screening, that in the opinion of the investigator and GSK Medical Monitor will interfere with the study or introduce additional safety risk to the subject.
* A serum sodium level =<125 milliequivalent (mEq) /liter (L) at screening
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within 56 days.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Unwillingness or inability to follow the procedures outlined in the protocol.

For Healthy Subjects (Cohort 2)

* ALT and bilirubin >1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Current or chronic history of liver disease (including acute or chronic Hepatitis B and C), or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
* QTc > 450 msec

NOTES:

The QTc is the QT interval corrected for heart rate according to Fridericia's formula (QTcF) machine-read or manually over-read.

For purposes of data analysis, QTcB, QTcF, or a composite of available values of QTc will be used as specified in the RAP.

* Systolic blood pressure outside the range of 90-145 mmHg, or diastolic blood pressure outside the range of 45-95mmHg or heart rate outside the range of 50-100 bpm for female subjects or 45-100 bpm for male subjects.
* Evidence of previous myocardial infarction or any clinically significant active cardiovascular disease that, in the opinion of the investigator, could interfere with the safety of the subject.
* Any clinically significant conduction abnormality (not including left or right complete bundle branch block) such as AV block [Mobitz type 2 second degree or higher AV block], Wolf Parkinson White [WPW] syndrome or other aberrant pathways.
* Sinus Pauses > 3 seconds.
* Any significant arrhythmia which, in the opinion of the principal investigator and GSK medical monitor, will interfere with the safety for the individual subject.
* Non-sustained or sustained ventricular tachycardia (>=3 consecutive ventricular ectopic beats).
* Signs of active infection that in the opinion of the investigator would interfere with the completion of study procedures or the safety of the subject.
* Fluctuating or deteriorating renal function or creatinine clearance (CLCR) < 90 mL/min (determined by 24-hour urine collection) at screening. Assessment of the stability of the subject's renal function will be determined by the investigator.
* Subjects with a pre-existing condition interfering with normal gastrointestinal anatomy or motility, hepatic and/or renal function, that could interfere with the absorption, metabolism, and/or excretion of the study drugs.
* History of inflammatory bowel disease.
* History of cholecystectomy or other gastrointestinal surgery (except appendectomy more than three months prior to study).
* History of peptic ulceration or pancreatitis within the preceding 6 months of screening.
* The use of any concurrent prohibited medications.
* History of regular alcohol consumption within 6 months of the study defined as:

An average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 g of alcohol: 12 ounces (360 mL) of beer, 5 ounces (150 mL) of wine or 1.5 ounces (45 mL) of 80 proof distilled spirits.

* A history of regular use of tobacco- or nicotine-containing products within 30 days prior to screening.
* Inability or unwillingness to comply with lifestyle and/or dietary restrictions
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation. In addition, if heparin is used during PK sampling, subjects with a history of sensitivity to heparin or heparin-induced thrombocytopenia should not be enrolled.
* Presence of hepatitis B surface antigen (or positive hepatitis B core antibody with negative hepatitis B surface antibody) or positive hepatitis C antibody test result at any time prior to first dose of study treatment.
* A pre-study screen positive for alcohol, cocaine, amphetamines, PCP, and/or barbiturates.
* A positive test for HIV antibody.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within 56 days.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Unwillingness or inability to follow the procedures outlined in the protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-07-13 (Actual); Primary Completion 2016-11-01 (Actual); Study Completion 2016-11-01 (Actual)

PRIMARY OUTCOMES:
Composite of PK parameters evaluated by measurement of AUC (0-infinity) and Cmax following single oral dose. | Samples will be collected at pre-dose (within 15 minutes prior to dose), 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 120 and 168 hours post dose.
  To compare effect of severe renal impairment on PK parameters for 744 assessed by Area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time (AUC[0-infinity]) and Maximum observed concentration (Cmax)

SECONDARY OUTCOMES:
Unbound concentration and unbound fraction in plasma of GSK1265744 at 2 and 24 hours post dose | Samples will be collected at 2 and 24 hours post dose.
  To evaluate impact of severe renal impairment on the plasma concentration of 744 assessed by measuring unbound concentration and unbound fraction in plasma of 744
Composite of PK parameters for GSK1265744 evaluated by measurement of Plasma AUC(0-t), %AUCex, C24, t1/2, CL/F, tlag, tmax and Vz/F following a single oral dose | Samples will be collected at pre-dose (within 15 minutes prior to dose), 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 120 and 168 hours post dose.
  To evaluate composite of PK parameters for 744 assessed by Area under the concentration-time curve from time zero (pre-dose) to the time of the last quantifiable concentration (AUC[0-t]), Percentage of AUC(0- infinity) obtained by extrapolation (%AUCex), Concentration observed 24-hours post dose (C24), Apparent terminal phase half-life (t1/2), Lag time before observation of drug concentrations in sampled matrix (tlag), Time of occurrence of Cmax (tmax), Apparent clearance following oral dosing (CL/F), apparent terminal phase volume of distribution (Vz/F)
Number of participants with adverse events as measure of safety and tolerability | Day -1 to Day 15
  To evaluate Safety and tolerability of single oral dose of 744 assessed by clinical safety data from number of participants with adverse event. Reporting of adverse event from the start of Study Treatment and until the final follow-up visit. Intensity of AEs will be categorized as mild, moderate or severe.
Safety and tolerability of single oral dose of 744 assessed by clinical laboratory tests | 14 Days
  To evaluate Safety and tolerability of single oral dose of 744 assessed by safety laboratory tests including Hematology, clinical chemistry, urinalysis and additional parameters
Safety and tolerability of single oral dose of 744 assessed by12-Lead electrocardiogram | 2 Days
  To evaluate Safety and tolerability of single oral dose of 744 assessed by12-Lead Electrocardiogram (ECG).
Safety and tolerability of single oral dose of 744 assessed by vital signs | 14 Days
  To evaluate Safety and tolerability of single oral dose of 744 assessed by vital signs. It will include temperature, systolic and diastolic blood pressure, pulse rate, and respiratory rate.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (2):
- United States (2):
  - GSK Investigational Site, Lakewood, Colorado
  - GSK Investigational Site, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=20362

REFERENCES:
- [Background] Parasrampuria R, Ford SL, Lou Y, Fu C, Bakshi KK, Tenorio AR, Trezza C, Spreen WR, Patel P. A Phase I Study to Evaluate the Pharmacokinetics and Safety of Cabotegravir in Adults With Severe Renal Impairment and Healthy Matched Control Participants. Clin Pharmacol Drug Dev. 2019 Jul;8(5):674-681. doi: 10.1002/cpdd.664. Epub 2019 Feb 27. PMID 30809978